CLINICAL TRIAL: NCT06741358
Title: Use of the Glialia Supplement in the Treatment of Persistent Perceptual Postural Imbalance: A Triple-Blind, Randomized, Placebo-Controlled Pilot Clinical Trial
Brief Title: Using Glialia for Treating Persistent Perceptual Postural Dizziness
Acronym: GLI-PPPD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N.153/SL/24
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: Persistent Postural Perceptual Dizziness
Keywords: Persistent Perceptual Postural Dizziness; Functional disorder; Neuroinflammation; Human Palmitoylethanolamide (umPEA); Neurofilaments; Balance
MeSH Terms: conditions — Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glialia (Experimental): Participants in the PPPD-Glialia group must be between the ages of 18 and 65 years and have a confirmed diagnosis of Persistent Perceptual Postural Dizziness (PPPD). They must also either have recovered from a COVID-19 infection or have no history of such an infection. Individuals with concurrent neurological or otological disorders, as well as pregnant women, will be excluded from this group.
  Interventions: Other: Glialia
- Placebo (Placebo Comparator): Participants in the PPPD-Glialia group must be between the ages of 18 and 65 years and have a confirmed diagnosis of Persistent Perceptual Postural Dizziness (PPPD). They must also either have recovered from a COVID-19 infection or have no history of such an infection. Individuals with concurrent neurological or otological disorders, as well as pregnant women, will be excluded from this group.
  Interventions: Other: Placebo
- Control group (Other): The Control Group will consist of individuals aged between 18 and 65 years who have a previous history of COVID-19 infection, matched for timing with the PPPD-Glialia group. Exclusion criteria for this group will also include the presence of any neurological or otological disorders and pregnancy, ensuring that the results are focused on the impact of the Glialia supplement in the context of PPPD and recovery from COVID-19.
  Interventions: Other: Control

INTERVENTIONS:
Other: Glialia — Participants in the PPPD-Glialia group will receive the Glialia supplement, which contains 700 mg of Palmitoylethanolamide (umPEA) along with 70 mg of additional supportive ingredients. Each participant will be instructed to take two soluble sachets daily for a total duration of 60 days. This group aims to evaluate the effects of Glialia on PPPD, with outcomes assessed for neuroinflammation, mental clarity, quality of life, balance, and gait quality.
  Arms: Glialia
Other: Placebo — Participants assigned to the PPPD-Placebo group will receive a placebo that is designed to be indistinguishable from the Glialia supplement in terms of appearance and packaging. They will also take two soluble sachets daily for 60 days. The purpose of this group is to serve as a control to evaluate the effects of the Glialia supplement by comparing the outcomes with those of the PPPD-Glialia group. The same assessments for neuroinflammation, mental clarity, quality of life, balance, and gait quality will be performed.
  Arms: Placebo
Other: Control — Individuals in the Control Group will receive the same Glialia supplement as the PPPD-Glialia group, containing 700 mg of Palmitoylethanolamide (umPEA) and 70 mg of supportive ingredients. They will also take two soluble sachets daily for 60 days. The primary goal for this group is to assess how the Glialia supplement affects neuroinflammation and related outcomes in individuals who have recovered from COVID-19 but do not have PPPD. This comparison will help clarify the potential effects of Glialia in the context of both PPPD and recovery from COVID-19.
  Arms: Control group

SUMMARY:
This pilot study will involve 30 participants recruited from the Santa Lucia Foundation IRCCS, including 20 patients diagnosed with Persistent Perceptual Postural Dizziness (PPPD), and might or might not have previously contracted Sars Cov2 infection. They who will be randomly assigned to receive either the Glialia supplement or placebo. Additionally, 10 control participants who have recovered from COVID-19 will receive Glialia to help assess the influence of previous COVID-19 infection on neuroinflammation levels. The study aims to compare baseline neuroinflammation levels between PPPD patients and controls, measure changes in neuroinflammation in all groups after treatment and to determine if the reduction in neuroinflammation is more significant in the Glialia group compared to the placebo group. The trial will be conducted in a triple-blind manner, ensuring that neither participants nor researchers know the treatment assignments. Each participant will receive sachets to be taken daily for 60 days, with the study providing both the Glialia supplement and placebo at no cost.

ELIGIBILITY:
Inclusion criteria for all groups:

-Age between 18 and 65 years.

Inclusion criteria for the PPPD-glialia group:

* Diagnosis of PPPD;
* Recovery from COVID-19 infection or absence of previous infection.

Inclusion criteria for the PPPD-placebo group:

* Diagnosis of PPPD;
* Recovery from COVID-19 infection or absence of previous infection (matched to the PPPD-glialia group).

Exclusion criteria for all PPPD-group:

* Presence of concurrent neurological and otological disorders other than PPPD;
* Pregnant women.

Inclusion criteria for the control group:

-Previous COVID-19 infection (matched for timing to the PPPD-glialia group).

Exclusion criteria for the control group:

* Presence of neurological and otological disorders;
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-21 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Neuroinflammation Assessment | T0 (Baseline); T1 (60 days)
  The neuroinflammation assessment will evaluate serum neurofilament light chain (NfL) levels as a biomarker for neuroinflammation in participants with PPPD and controls. Blood samples will be collected via venipuncture at the Foundation Santa Lucia IRCCS. The analysis will utilize a sensitive enzyme-linked immunosorbent assay (ELISA) method to quantify NfL levels. The Simoa NF-Light advantage kit will enable accurate detection of low concentrations. This assessment aims to compare neuroinflammation levels at baseline (T0) and after treatment (T1) across the study groups.

SECONDARY OUTCOMES:
Gait Quality Assessment | T0 (Baseline); T1 (60 days)
  Gait quality will be assessed using inertial sensors. Set of magneto-inertial sensors (Opal, APDM Inc., Portland, Oregon, USA) will be used during the execution of walking motor tasks. Changes of continuous accelerometer signals will be recorded.
Video Head Impulse Test (vHIT) | T0 (Baseline).
  The Video Head Impulse Test (vHIT) is performed to assess the vestibulo-ocular reflex (VOR). Conducted before T0, this test ensures that participants do not have underlying VOR dysfunction prior to inclusion in the study.
Dizziness Handicap Inventory (DHI) | T0 (Baseline); T1 (60 days)
  The Dizziness Handicap Inventory (DHI) measures the impact of dizziness on an individual's daily life and activities. Participants will complete this questionnaire at T0 and T1 to assess any changes in disability related to dizziness. The DHI provides insights into the physical, emotional, and functional limitations experienced by patients, facilitating a comprehensive evaluation of the treatment's effectiveness in improving quality of life. The maximum score for the DHI ranges from 0 to 100, with higher scores indicating greater instability.
Niigata Questionnaire | T0 (Baseline); T1 (60 days)
  The Niigata questionnaire assesses subjective symptoms related to PPPD. It is administered to participants at both T0 and T1 to evaluate changes in symptom perception over the treatment period. The questionnaire consists of various items that help quantify the intensity and frequency of PPPD symptoms, allowing for a comparative analysis of symptom improvement in the PPPD-glialia and PPPD-placebo groups. The maximum score is 72, with higher scores reflecting greater instability. Each of its three domains (upright posture/walking, movement, and visual stimulation) has a maximum score of 24.
Brain Fog Scale (BFS) | T0 (Baseline); T1 (60 days)
  The Brain Fog Scale (BFS) is designed to evaluate cognitive clarity and mental processing in participants. Administered at both T0 and T1, this scale focuses on self-reported cognitive difficulties, such as concentration, memory, and mental fatigue. Changes in BFS scores will help determine the cognitive effects of the treatment, particularly in the context of PPPD-related cognitive symptoms.
Personality Traits Assessment (NEO-P-I-3) | T0 (Baseline)
  The NEO-P-I-3 questionnaire will be administered at T0 to evaluate personality traits, particularly focusing on neuroticism, which is relevant for understanding the psychological aspects of PPPD. This assessment will provide baseline data on individual personality profiles and allow for exploration of potential correlations between personality traits and treatment outcomes in PPPD patients. A statistical analysis will be conducted to evaluate specific areas of personality traits.

CONTACTS AND LOCATIONS:
Overall Officials: Iole Indovina, PhD, Principal Investigator — Department of Systems Medicine, University of Rome Tor Vergata Rome, Italy ; Centre of Space Bio-medicine, University of Rome Tor Vergata Rome, Italy ; Laboratory of Neuromotor Physiology, IRCCS Santa Lucia Foundation Rome, Italy.; Arianna Di Stadio, PhD, Study Director — GF Ingrassia Department, University of Catania, Catania, Italy.; Diego Piatti, PT, Study Chair — Laboratory of Neuromotor Physiology, IRCCS Santa Lucia Foundation, 00179 Rome, Italy.; Gianluca Paolocci, PhD, Study Chair — Department of Biomedical and Dental Sciences and Morphofunctional Imaging, University of Messina, 98125 Messina, Italy; Laboratory of Neuromotor Physiology, IRCCS Santa Lucia Foundation, 00179 Rome, Italy.; Gianfranco Bosco, PhD, Study Chair — Department of Systems Medicine, University of Rome Tor Vergata Rome, Italy ; Centre of Space Bio-medicine, University of Rome Tor Vergata Rome, Italy Laboratory of Neuromotor Physiology, IRCCS Santa Lucia Foundation Rome, Italy.; Cinzia Ciccacci, PhD, Study Chair — Unicamillus, Saint Camillus International University of Medical Sciences.; Marco Tramontano, PhD, Study Chair — Department of Biomedical and Neuromotor Sciences (DIBINEM), Alma Mater University of Bologna, 40138 Bologna, Italy; Unit of Occupational Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna, 40138 Bologna, Italy.; Francesca Giansanti, MSc, Study Chair — Unicamillus, Saint Camillus International University of Medical Sciences.
Locations (1):
- Fondazione Santa Lucia IRCCS, Rome, RM, Italy

REFERENCES:
- [Background] Tramontano M, Casagrande Conti L, Orejel Bustos AS, Ferri N, Lelli T, Nocentini U, Grasso MG, Turolla A, Pillastrini P, Manzari L. Abnormal Vestibulo-Ocular Reflex Function Correlates with Balance and Gait Impairment in People with Multiple Sclerosis. Audiol Res. 2024 Sep 9;14(5):799-808. doi: 10.3390/audiolres14050067. PMID 39311220
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Castillejos-Carrasco-Munoz R, Peinado-Rubia AB, Lerida-Ortega MA, Ibanez-Vera AJ, Tapia-Toca MC, Lomas-Vega R. Validity and reliability of the Niigata PPPD Questionnaire in a Western population. Eur Arch Otorhinolaryngol. 2023 Dec;280(12):5267-5276. doi: 10.1007/s00405-023-08038-1. Epub 2023 Jun 2. PMID 37266755
- [Background] Indovina I, Riccelli R, Staab JP, Lacquaniti F, Passamonti L. Personality traits modulate subcortical and cortical vestibular and anxiety responses to sound-evoked otolithic receptor stimulation. J Psychosom Res. 2014 Nov;77(5):391-400. doi: 10.1016/j.jpsychores.2014.09.005. Epub 2014 Sep 16. PMID 25262497